CLINICAL TRIAL: NCT01032694
Title: Non-Interventional Open Label Prospective Observational Comparative Study On Evaluation Of Compliance Of The Empiric Treatment With Azithromycin SR Versus Amoxiclav 1000 Mg In Adult Patients With Mild To Moderate Community Acquired Pneumonia
Acronym: PROSTO
Status: Terminated | Type: Observational
Why Stopped: This study was terminated January 11, 2011 due to low enrollment. This study is not being terminated because of safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0661200
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-11

CONDITIONS: Community-Acquired Pneumonia
Keywords: Community-Acquired Pneumonia; Azithromycin SR; Amoxiclav
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Z-max treated group: Patients with Community-Acquired Pneumonia
  Interventions: Drug: Azithromycin SR
- Amoxiclav treated group: Patients with Community-Acquired Pneumonia
  Interventions: Drug: Amoxiclav

INTERVENTIONS:
Drug: Azithromycin SR — Azithromycin SR, 2.0 g PO x 1 dose for treatment period
  Groups: Z-max treated group
Drug: Amoxiclav — Amoxiclav 1000 x twice daily, 10 days duration
  Groups: Amoxiclav treated group

SUMMARY:
To compare compliance between patients with CAP treated with Azithromycin SR 2.0 g single dose orally and those treated with Amoxiclav - 1000 mg twice daily 10 days for the empiric treatment of CAP in outpatient clinic practice.

ELIGIBILITY:
Inclusion Criteria:

* Males or not pregnant or lactating females, 18 years of age or older, for whom oral antibacterial therapy is indicated with clinically evidence of Diagnosis of pneumonia, based on usual clinical practice:

  1. Physical examination and auscultatory findings (dullness on percussion, bronchial breath sounds, egophony, dry or fine most rales).
  2. Body temperature >38 degrees C.

Exclusion Criteria:

* Known or suspected hypersensitivity or intolerance or contraindications to Azithromycin.
* Amoxiclav according to LPDs, pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Community-Acquired Pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661200&StudyName=Non-Interventional%20Open%20Label%20Prospective%20Observational%20Comparative%20Study%20On%20Evaluation%20Of%20Compliance%20Of%20The%20Empiric%20Treatment%20With%20Azithromyc

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: A single dose of azithromycin 2000 milligram (mg) sustained release (SR) tablet administered orally.
- Amoxiclav: Amoxiclav 1000 mg tablet administered twice daily (BID) orally for 10 days.
Period: Overall Study
Arm/Group | Azithromycin | Amoxiclav
Started | 20 | 10
Completed | 20 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Amoxiclav | Total
Number analyzed (Participants) | 20 | 10 | 30
Age Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (18.0) | 40.1 (7.9) | 43.9 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response of Very Convenient or Somewhat Convenient
Description: Participant reported outcome questionnaire was the assessment of participant's convenience with drug treatment based on following categories: very convenient or somewhat convenient and not convenient or not at all convenient. Value of 1 was reported if participant answered 'very convenient' or 'somewhat convenient' and 0 if participant answered 'not convenient' or 'not at all convenient'.
Time Frame: Days 11-12
Population: The Full Analysis Set (FAS) population included all participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy evaluation. Missing observations were not imputed. 'N' signifies the number of participants with non-missing data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Azithromycin | Amoxiclav
Number analyzed (Participants) | 19 | 6
Percentage of Participants | 100 | 100

2. Secondary Outcome: Percent Compliance With the Prescribed Treatment Regimen
Description: Percent compliance with the prescribed treatment regimen was calculated as 100 multiplied by (number of tablets taken by the participant divided by number of tablets prescribed).
Time Frame: Days 11-12
Population: The FAS population included all participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Percent compliance
Arm/Group | Azithromycin | Amoxiclav
Number analyzed (Participants) | 20 | 10
Percent compliance | 100.0 (0.0) | 100.0 (0.0)

3. Secondary Outcome: Percentage of Participants Who Were 100 Percent Compliant With Prescribed Treatment Regimen
Description: Percent compliance with the prescribed treatment regimen was calculated as 100 multiplied by (number of tablets taken by the participant divided by number of tablets prescribed). Value of 1 was reported if percent compliance equals to 100, and 0 if percent compliance was non-missing and less than 100.
Time Frame: Days 11-12
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Azithromycin | Amoxiclav
Number analyzed (Participants) | 20 | 10
Percentage of Participants | 100 | 100

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Azithromycin | Amoxiclav
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 2/20 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=20) | Amoxiclav (N=10)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.